CLINICAL TRIAL: NCT06919484
Title: The Physiological Effect of RCexp on Ventilation/Perfusion Distribution in Patients With ARDS
Brief Title: The Physiological Effect of RCexp on Ventilation/Perfusion Distribution
Status: Recruiting | Type: Observational
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, PhD, Southeast University, China
Other Study IDs: RCexp_ventilation/perfusion
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Acute Respiratory Distress Syndrome; Mechanical Ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- mechanically ventilated patients with ARDS
  Interventions: Other: RCexp

INTERVENTIONS:
Other: RCexp — patients received different RCexp

SUMMARY:
With the exception of setting the positive end-expiratory pressure (PEEP), the expiratory phase is commonly overlooked during MV. The expiratory time constant (RCexp) plays an important role in understanding the mechanical properties of the respiratory system in patients receiving mechanical ventilation. However, it is unclear that the effect of expiratory time constant on the ventilation and perfusion distribution.

DETAILED DESCRIPTION:
With the exception of setting the positive end-expiratory pressure (PEEP), the expiratory phase is commonly overlooked during MV. The expiratory time constant (RCexp) plays an important role in understanding the mechanical properties of the respiratory system in patients receiving mechanical ventilation. However, it is unclear that the effect of expiratory time constant on the ventilation and perfusion distribution.

ELIGIBILITY:
Inclusion Criteria:

adult patients with ARDS receiving mechanical ventilation no more than 72 hours

Exclusion Criteria:

1. age <18 years old
2. patient undergoing legal protection
3. contra-indications to EIT (e. g. severe chest trauma or wounds)
4. pneumothorax
5. patient undergoing ECMO
6. pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Intubated patients with moderate and severe ARDS (Berlin definition, PaO2/FiO2 ≤200 mmHg at PEEP 5 cmH2O)
  2. undergoing deep sedation on controlled mechanical ventilation within72 hours after ARDS onset
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in ventilation/perfusion mismatch | 4 hours
  ventilation/perfusion mismatch is measured by EIT

SECONDARY OUTCOMES:
Difference in dead space | 4 hours
  dead space is measured by EIT
Difference in shunt | 4 hours
  shunt is measured by EIT

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital, School of Medicine, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No